CLINICAL TRIAL: NCT05759000
Title: The Effect of Early Inpatient Initiation of Dapagliflozin on the Health-related Quality of Life of Patients With Heart Failure With All Range of Ejection Fraction: a Local Registry
Brief Title: Dapa Acute Heart Failure Study
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.501
Record Dates: First submitted 2022-10-13; First posted 2023-03-08 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: Dapagliflozin; acute heart failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dapagliflozin — Sodium-glucose cotransporter-2 (SGLT2) inhibitor is considered one of the four foundational therapies (ACE-I or ARNI, beta-blockers, MRA, and SGLT2 inhibitors) for HFrEF (6). However, guidelines do not specify the sequence and the timing of which therapy to be commenced. In particular, dapagliflozin has been shown in randomized controlled trials to reduce the combined risk of cardiovascular death or HF hospitalization and improve quality of life in HF patients with both reduced ejection fraction (HFrEF) and preserved ejection fraction (HFpEF), respectively, regardless of the presence or absence of diabetes in the DAPA-HF and DELIVER trials (

SUMMARY:
Heart failure (HF) is one of the most important reasons for hospital admission and is associated with high mortality and morbidity. After discharge, up to 40% of patients are readmitted within 6 months and 1-year post-discharge mortality is high. The cost burden of treating patients with HF is high and ~80% of healthcare costs are related to hospital admissions.

Sodium-glucose cotransporter-2 (SGLT2) inhibitor is considered one of the four foundational therapies (ACE-I or ARNI, beta-blockers, MRA, and SGLT2 inhibitors) for HFrEF.

This is an investigator-initiated, prospective, single-centre, registry that evaluates the change in HRQL as measured by the KCCQ-TSS after the initiation of Dapagliflozin.

DETAILED DESCRIPTION:
Heart failure (HF) is one of the most important reasons for hospital admission and is associated with high mortality and morbidity and poor quality of life (1). After discharge, up to 40% of patients are readmitted within 6 months and 1-year post-discharge mortality is high (2-4). The cost burden of treating patients with HF is high and ~80% of healthcare costs are related to hospital admissions (5).

Sodium-glucose cotransporter-2 (SGLT2) inhibitor is considered one of the four foundational therapies (ACE-I or ARNI, beta-blockers, MRA, and SGLT2 inhibitors) for HFrEF (6) However, guidelines do not specify the sequence and the timing of which therapy to be commenced. In particular, dapagliflozin has been shown in randomized controlled trials to reduce the combined risk of cardiovascular death or HF hospitalization and improve quality of life in HF patients with both reduced ejection fraction (HFrEF) and preserved ejection fraction (HFpEF), respectively, regardless of the presence or absence of diabetes in the DAPA-HF and PRESERVED-HF trials (7, 8).

HF patient usually has poor QoL, and health-related quality of life (HRQL) measure has been shown to be associated with all cause death and HF hospitalization in a multinational study (9). There exist a geographical and ethnical variation in patients HRQL and clinical outcomes amongst various countries (9). The Kansas City Cardiomyopathy Questionnaire-total symptom scores (KCCQ-TSS) is a simple, widely available, and inexpensive tool that characterizes a patient's HF-related health status. Showing that it can be used as a marker to predict major clinical outcomes in a wide spectrum of patients with HF across the world would confirm its usefulness in research as well as in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age >18 hospitalized for primary diagnosis of acute HF
2. Dyspnoea (exertional or at rest) and 1 of the following signs:

   * Congestion on chest X-ray
   * Rales on chest auscultation
   * Clinically relevant oedema (e.g. ≥1+ on a 0 to 3+ scale)
   * Elevated jugular venous pressure
3. NT-proBNP ≥300 ng/L (If ongoing atrial fibrillation/flutter at recruitment, NT-pro BNP must be ≥ 600 pg/mL.4. 5).

Exclusion Criteria:

1. Cardiogenic shock
2. Current hospitalization for acute HF primarily triggered by pulmonary embolism or cerebrovascular accident.
3. Interventions in the past 30 days prior or planned during the study: Major cardiac surgery, or TAVI, or PCI, or MitraClip
4. Current or expected heart transplant, LVAD, on IABP or other forms of mechanical support.
5. Haemodynamically severe uncorrected primary cardiac valvular disease planned for surgery or intervention during the course of the study.
6. eGFR <20 mL/min/1.73m2 as measured during index hospitalization (latest measurement before randomization) or patients requiring dialysis
7. Type 1 diabetes mellitus
8. History of ketoacidosis, including diabetic ketoacidosis
9. Prior treatment with SGLT2 inhibitors in 90 days prior to current admission.
10. Documented severe allergy or intolerance to SGLT2 inhibitors.
11. Pregnant subjects

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is based on the primary objective and calculation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2025-09-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in KCCQ-TSS | Change from baseline in KCCQ-TSS after 90 days of treatment.

SECONDARY OUTCOMES:
Change from baseline in log-transformed NT-proBNP level | Change from baseline in log-transformed NT-proBNP level over 90 days of treatment
Change in NYHA class | Change in NYHA class over 90 days of treatment
Days alive and out of hospital from study drug initiation | 90 days
Days alive and out of hospital from study drug initiation | Days alive and out of hospital from study drug initiation until 90 days after randomization
Time to first occurrence of cardiovascular death or heart Dapa AHF study Ver. 1.4 dated 7Oct2022 2 failure event | 90 days
Occurrence of HHF | Occurrence of HHF until 90 days after initial hospital discharge
Occurrence of Sustained eGFR reduction of ≥40% eGFR, or - Sustained eGFR <15mL/min/1.73m2 for patients with baseline eGFR ≥30 mL/min/1.73m2 - Sustained eGFR <10mL/min/1.73m2 for patients with baseline eGFR <30 mL/min/1.73m2. | Occurrence of Sustained eGFR until 90 days after initial hospital discharge
Change from baseline in 6MWD | Change from baseline in 6MWD at 90 days
Cost effectiveness of early initiation of dapagliflozin for heart failure events avoided | 90 days
Clinical benefit | 90 days
  a composite of all-cause mortality, number of heart failure events (including hospitalization for HFs, urgent heart failure visits and unplanned outpatient visits)
quality-of-life years (QALY) gained of dapagliflozin for heart failure events avoided | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Result] Krumholz HM, Merrill AR, Schone EM, Schreiner GC, Chen J, Bradley EH, Wang Y, Wang Y, Lin Z, Straube BM, Rapp MT, Normand SL, Drye EE. Patterns of hospital performance in acute myocardial infarction and heart failure 30-day mortality and readmission. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):407-13. doi: 10.1161/CIRCOUTCOMES.109.883256. Epub 2009 Jul 9. PMID 20031870
- [Result] Chun S, Tu JV, Wijeysundera HC, Austin PC, Wang X, Levy D, Lee DS. Lifetime analysis of hospitalizations and survival of patients newly admitted with heart failure. Circ Heart Fail. 2012 Jul 1;5(4):414-21. doi: 10.1161/CIRCHEARTFAILURE.111.964791. Epub 2012 May 2. PMID 22556322
- [Result] Joynt KE, Jha AK. Who has higher readmission rates for heart failure, and why? Implications for efforts to improve care using financial incentives. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):53-9. doi: 10.1161/CIRCOUTCOMES.110.950964. Epub 2010 Dec 14. PMID 21156879
- [Result] Braunschweig F, Cowie MR, Auricchio A. What are the costs of heart failure? Europace. 2011 May;13 Suppl 2:ii13-7. doi: 10.1093/europace/eur081. PMID 21518742
- [Result] Writing Committee; Maddox TM, Januzzi JL Jr, Allen LA, Breathett K, Butler J, Davis LL, Fonarow GC, Ibrahim NE, Lindenfeld J, Masoudi FA, Motiwala SR, Oliveros E, Patterson JH, Walsh MN, Wasserman A, Yancy CW, Youmans QR. 2021 Update to the 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment: Answers to 10 Pivotal Issues About Heart Failure With Reduced Ejection Fraction: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2021 Feb 16;77(6):772-810. doi: 10.1016/j.jacc.2020.11.022. Epub 2021 Jan 11. No abstract available. PMID 33446410
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Result] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Result] Johansson I, Joseph P, Balasubramanian K, McMurray JJV, Lund LH, Ezekowitz JA, Kamath D, Alhabib K, Bayes-Genis A, Budaj A, Dans ALL, Dzudie A, Probstfield JL, Fox KAA, Karaye KM, Makubi A, Fukakusa B, Teo K, Temizhan A, Wittlinger T, Maggioni AP, Lanas F, Lopez-Jaramillo P, Silva-Cardoso J, Sliwa K, Dokainish H, Grinvalds A, McCready T, Yusuf S; G-CHF Investigators. Health-Related Quality of Life and Mortality in Heart Failure: The Global Congestive Heart Failure Study of 23 000 Patients From 40 Countries. Circulation. 2021 Jun;143(22):2129-2142. doi: 10.1161/CIRCULATIONAHA.120.050850. Epub 2021 Apr 28. PMID 33906372